CLINICAL TRIAL: NCT02711345
Title: A Phase I Dose Finding Study of Oral LTT462 in Adult Patients With Advanced Solid Tumors Harboring MAPK Pathway Alterations.
Brief Title: A Phase I Clinical Study With Investigational Compound LTT462 in Adult Patients With Specific Advanced Cancers.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: considering the limited clinical activity observed with LTT462, the decision was made to not open the dose expansion phase of the study
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLTT462X2101; 2015-003614-24 (EudraCT Number)
Record Dates: First submitted 2016-02-16; First posted 2016-03-17 (Estimated); Results first posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-08

CONDITIONS: Ovarian Neoplasms; Non-Small-Cell Lung Carcinoma; Melanoma; Other Solid Tumors
Keywords: LTT462; ERK; MAPK; solid tumor
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Escalation (Experimental)
  Interventions: Drug: LTT462
- Expansion Group 1 (Experimental)
  Interventions: Drug: LTT462
- Expansion Group 2 (Experimental)
  Interventions: Drug: LTT462
- Expansion Group 3 (Experimental)
  Interventions: Drug: LTT462
- Expansion Group 4 (Experimental)
  Interventions: Drug: LTT462

INTERVENTIONS:
Drug: LTT462 — ERK Inhibitor

SUMMARY:
A phase I study of LTT462 in patients with advanced solid tumors that harbor MAPK pathway alterations.

ELIGIBILITY:
Inclusion Criteria:

* Patient (male or female) ≥12 years of age
* ECOG (Eastern Cooperative Oncology Group) performance status ≤1
* Must have progressed following standard therapy, or for whom, in the opinion of the Investigator, no effective standard therapy exists, is tolerated or appropriate.
* Patients must be willing and able to undergo study required biopsies.
* Presence of at least one measurable lesion according to RECIST v1.1.
* Documented MAPK pathway alteration

Exclusion Criteria:

* Prior treatment with ERK inhibitors.
* History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO.
* Any medical condition that would, in the investigator's judgment, prevent the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures.
* Patients receiving proton pump inhibitors (PPI) which cannot be discontinued 3 days prior to the start study treatment and for the duration of the study.
* Patients with malignant disease other than that being treated in the study.
* Clinically significant cardiac disease.

Other protocol-defined exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-04-15 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- United States (2):
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Houston, Texas
- Novartis Investigative Site, Essen, Germany
- Novartis Investigative Site, Chuo Ku, Tokyo, Japan
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- Novartis Investigative Site, Bellinzona, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- LTT462 45 mg QD: Participants received LTT462 45 milligram (mg) once daily (QD)
- LTT462 100 mg QD: Participants received 100 mg LTT462 QD as oral capsules.
- LTT462 150 mg QD: Participants received 150 mg LTT462 QD as oral capsules.
- LTT462 200 mg QD: Participants received 200 mg LTT462 QD as oral capsules.
- LTT462 300 mg QD: Participants received 300 mg LTT462 QD as oral capsules.
- LTT462 400 mg QD: Participants received 400 mg LTT462 QD as oral capsules.
- LTT462 450 mg QD: Participants received 450 mg LTT462 QD as oral capsules.
- LTT462 600 mg QD: Participants received 600 mg LTT462 QD as oral capsules.
- LTT462 150 mg BID: Participants received 150 mg LTT462 twice daily (BID) as oral capsules.
- LTT462 200 mg BID: Participants received 200 mg LTT462 BID as oral capsules.
Period: Overall Study
Arm/Group | LTT462 45 mg QD | LTT462 100 mg QD | LTT462 150 mg QD | LTT462 200 mg QD | LTT462 300 mg QD | LTT462 400 mg QD | LTT462 450 mg QD | LTT462 600 mg QD | LTT462 150 mg BID | LTT462 200 mg BID
Started | 2 | 3 | 6 | 4 | 8 | 6 | 12 | 6 | 6 | 12
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 3 | 6 | 4 | 8 | 6 | 12 | 6 | 6 | 12
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Progressive disease | 1 | 3 | 5 | 3 | 7 | 2 | 8 | 4 | 5 | 6
Not completed — Subject/guardian decision | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 0 | 4
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- LTT462 45 mg QD: Participants received 45 mg LTT462 once QD as oral capsules.
- LTT462 150 mg BID: Participants received 150 mg LTT462 BID as oral capsules.
- Total: Total of all reporting groups
Arm/Group | LTT462 45 mg QD | LTT462 100 mg QD | LTT462 150 mg QD | LTT462 200 mg QD | LTT462 300 mg QD | LTT462 400 mg QD | LTT462 450 mg QD | LTT462 600 mg QD | LTT462 150 mg BID | LTT462 200 mg BID | Total
Number analyzed (Participants) | 2 | 3 | 6 | 4 | 8 | 6 | 12 | 6 | 6 | 12 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Between 18 and 65 years | 1 | 2 | 5 | 3 | 5 | 5 | 7 | 5 | 5 | 6 | 44
  >=65 years | 1 | 1 | 1 | 1 | 2 | 1 | 5 | 1 | 1 | 6 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4 | 2 | 6 | 4 | 5 | 4 | 4 | 7 | 40
  Male | 1 | 0 | 2 | 2 | 2 | 2 | 7 | 2 | 2 | 5 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 1 | 2 | 5 | 2 | 6 | 2 | 7 | 4 | 5 | 8 | 42
  Black | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3
  Asian | 1 | 1 | 1 | 1 | 1 | 3 | 4 | 0 | 0 | 2 | 14
  Unknown | 00 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An adverse events is defined as the appearance of (or worsening of any pre-existing) undesirable signs, symptoms, or medical conditions that occur after participant's signed informed consent has been obtained. A SAE is described as any adverse event that leads to death, is life threatening, causes or prolongs hospitalization, results in a congenital anomaly, or any other important medical event not described above.
Time Frame: Up to 2.8 years
Population: The safety set included all participants who had received at least one dose of LTT462.
Measure: Number; unit: Percentage of participants
Groups:
- LTT462 45 mg QD: Participants received 45 mg LTT462 QD as oral capsules.
Arm/Group | LTT462 45 mg QD | LTT462 100 mg QD | LTT462 150 mg QD | LTT462 200 mg QD | LTT462 300 mg QD | LTT462 400 mg QD | LTT462 450 mg QD | LTT462 600 mg QD | LTT462 150 mg BID | LTT462 200 mg BID
Number analyzed (Participants) | 2 | 3 | 6 | 4 | 8 | 6 | 12 | 6 | 6 | 12
Percentage of participants
  AEs | 2 | 3 | 6 | 4 | 8 | 6 | 12 | 5 | 6 | 12
  SAEs | 1 | 0 | 3 | 1 | 5 | 1 | 8 | 4 | 3 | 5

2. Primary Outcome: Percentage of Participants With Dose Limiting Toxicities (DLTs)
Description: Percentage of participants with dose limiting toxicity were reported.
Time Frame: Up to 2.8 years
Population: The dose determining set included all participants from the safety set enrolled in the escalation part of the study who, during the first 28 days of dosing, had received at least 75 percent of the planned daily doses of LTT462 and had had sufficient safety evaluations, or had experienced a DLT.
Measure: Number; unit: Percentage of participants
Arm/Group | LTT462 45 mg QD | LTT462 100 mg QD | LTT462 150 mg QD | LTT462 200 mg QD | LTT462 300 mg QD | LTT462 400 mg QD | LTT462 450 mg QD | LTT462 600 mg QD | LTT462 150 mg BID | LTT462 200 mg BID
Number analyzed (Participants) | 2 | 3 | 6 | 4 | 7 | 4 | 7 | 3 | 4 | 9
Percentage of participants | 0 | 0 | 16.7 | 25.0 | 0 | 0 | 28.6 | 100 | 0 | 44.4

3. Primary Outcome: Percentage of Participants With at Least One Dose Reduction
Description: Percentage of participants with at least one dose reduction were reported.
Time Frame: Up to 2.8 years
Population: The safety set included all participants who had received at least one dose of LTT462.
Measure: Number; unit: Percentage of participants
Arm/Group | LTT462 45 mg QD | LTT462 100 mg QD | LTT462 150 mg QD | LTT462 200 mg QD | LTT462 300 mg QD | LTT462 400 mg QD | LTT462 450 mg QD | LTT462 600 mg QD | LTT462 150 mg BID | LTT462 200 mg BID
Number analyzed (Participants) | 2 | 3 | 6 | 4 | 8 | 6 | 12 | 6 | 6 | 12
Percentage of participants | 0 | 0 | 16.7 | 0 | 0 | 0 | 16.7 | 33.3 | 16.7 | 33.3

4. Primary Outcome: Percentage of Participants With at Least One Dose Interruptions
Description: Percentage of participants with at least dose interruptions were reported.
Time Frame: Up to 2.8 years
Population: The safety set included all participants who had received at least one dose of LTT462.
Measure: Number; unit: Percentage of participants
Arm/Group | LTT462 45 mg QD | LTT462 100 mg QD | LTT462 150 mg QD | LTT462 200 mg QD | LTT462 300 mg QD | LTT462 400 mg QD | LTT462 450 mg QD | LTT462 600 mg QD | LTT462 150 mg BID | LTT462 200 mg BID
Number analyzed (Participants) | 2 | 3 | 6 | 4 | 8 | 6 | 12 | 6 | 6 | 12
Percentage of participants | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100

5. Primary Outcome: Dose Intensity Received by Participants
Description: Dose intensity of LTT462 received by treatment group was reported.
Time Frame: Up to 2.8 years
Population: The safety set included all participants who had received at least one dose of LTT462.
Measure: Mean (Standard Deviation); unit: milligram per day (mg/day)
Arm/Group | LTT462 45 mg QD | LTT462 100 mg QD | LTT462 150 mg QD | LTT462 200 mg QD | LTT462 300 mg QD | LTT462 400 mg QD | LTT462 450 mg QD | LTT462 600 mg QD | LTT462 150 mg BID | LTT462 200 mg BID
Number analyzed (Participants) | 2 | 3 | 6 | 4 | 8 | 6 | 12 | 6 | 6 | 12
milligram per day (mg/day) | 65.3 (28.74) | 98.1 (3.21) | 133.9 (21.84) | 200.0 (0.00) | 272.7 (30.90) | 326.7 (81.54) | 409.2 (64.88) | 468.2 (171.48) | 131.6 (22.08) | 178.0 (35.32)

6. Secondary Outcome: Percentage of Participants With Overall Response Rate (ORR)
Description: Percentage of participants with overall response rate were reported.
Time Frame: Every 2 cycles after starting LTT462 treatment until end of treatment (Up to 2.8 years)
Population: The full analysis set included all participants who had received at least one dose of LTT462.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LTT462 45 mg QD | LTT462 100 mg QD | LTT462 150 mg QD | LTT462 200 mg QD | LTT462 300 mg QD | LTT462 400 mg QD | LTT462 450 mg QD | LTT462 600 mg QD | LTT462 150 mg BID | LTT462 200 mg BID
Number analyzed (Participants) | 2 | 3 | 6 | 4 | 8 | 6 | 12 | 6 | 6 | 12
Percentage of participants | 0 [0 to 84.2] | 0 [0 to 70.8] | 0 [0 to 45.9] | 0 [0 to 60.2] | 0 [0 to 36.9] | 0 [0 to 45.9] | 0 [0 to 26.5] | 0 [0 to 45.9] | 0 [0 to 45.9] | 0 [0 to 26.5]

7. Secondary Outcome: Percentage of Participants With Disease Control Rate (DCR)
Description: Percentage of participants with disease control rate were reported.
Time Frame: Every 2 cycles after starting LTT462 treatment until end of treatment (Up to 2.8 years)
Population: The full analysis set included all participants who had received at least one dose of LTT462.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LTT462 45 mg QD | LTT462 100 mg QD | LTT462 150 mg QD | LTT462 200 mg QD | LTT462 300 mg QD | LTT462 400 mg QD | LTT462 450 mg QD | LTT462 600 mg QD | LTT462 150 mg BID | LTT462 200 mg BID
Number analyzed (Participants) | 2 | 3 | 6 | 4 | 8 | 6 | 12 | 6 | 6 | 12
Percentage of participants | 50.0 [1.3 to 98.7] | 0 [0 to 70.8] | 0 [0 to 45.9] | 0 [0 to 60.2] | 37.5 [8.5 to 75.5] | 16.7 [0.4 to 64.1] | 8.3 [0.2 to 38.5] | 16.7 [0.4 to 64.1] | 16.7 [0.4 to 64.1] | 0 [0 to 26.5]

8. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time between the date of the first documented response (complete response [CR] or partial response [PR]) and the date of progression.
Time Frame: Every 2 cycles after starting LTT462 treatment until end of treatment (Up to 2.8 years)
Population: As there were no participant achieving response (CR or PR) during escalation phase of the study (only stable disease was achieved). Therefore the evaluation of duration of response could not be performed.
Arm/Group | LTT462 45 mg QD | LTT462 100 mg QD | LTT462 150 mg QD | LTT462 200 mg QD | LTT462 300 mg QD | LTT462 400 mg QD | LTT462 450 mg QD | LTT462 600 mg QD | LTT462 150 mg BID | LTT462 200 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Progression Free Survival (PFS)
Description: Median time for progression free survival was reported.
Time Frame: Every 2 cycles after starting LTT462 treatment until end of treatment (Up to 2.8 years)
Population: The full analysis set included all participants who had received at least one dose of LTT462.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LTT462 45 mg QD | LTT462 100 mg QD | LTT462 150 mg QD | LTT462 200 mg QD | LTT462 300 mg QD | LTT462 400 mg QD | LTT462 450 mg QD | LTT462 600 mg QD | LTT462 150 mg BID | LTT462 200 mg BID
Number analyzed (Participants) | 2 | 3 | 6 | 4 | 8 | 6 | 12 | 6 | 6 | 12
months | 5.3 [1.3 to 9.2] | 1.6 [0.9 to 1.7] | 1.7 [1.2 to 2.0] | 1.9 [1.7 to 1.9] | 1.8 [1.2 to 5.1] | 2.1 [0.8 to 3.2] | 0.9 [0.8 to 1.6] | 1.4 [0.7 to 4.0] | 1.5 [1.2 to 3.7] | 1.6 [0.8 to 1.7]

10. Secondary Outcome: Overall Survival (OS) - Only for Dose Expansion Phase
Description: Median time for overall survival, only for dose expansion phase was reported.
Time Frame: Every 2 cycles after starting LTT462 treatment until end of treatment (Up to 2.8 years)
Population: Overall survival was not evaluated because the study ended before enrolling into the dose-expansion part.
Arm/Group | LTT462 45 mg QD | LTT462 100 mg QD | LTT462 150 mg QD | LTT462 200 mg QD | LTT462 300 mg QD | LTT462 400 mg QD | LTT462 450 mg QD | LTT462 600 mg QD | LTT462 150 mg BID | LTT462 200 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: The Maximum (Peak) Observed Plasma, Blood, Serum, or Other Body Fluid Drug Concentration (Cmax) After Single Dose Administration of LTT462
Description: Cmax is the maximum (peak) observed plasma, blood, serum, or other body fluid drug concentration after single dose administration expressed in mass x volume-1.
Time Frame: day 1, day 15
Population: Pharmacokinetic (PK) analysis set (PAS) included of all participants who have at least 1 PK blood sample providing measurable LTT462 and received at least 1 dose of study drug, didn't vomit within 4 hours postdose, had at least 1 primary PK parameter. Here 'n' number analyzed signifies number of participants who were evaluable at each time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | LTT462 45 mg QD | LTT462 100 mg QD | LTT462 150 mg QD | LTT462 200 mg QD | LTT462 300 mg QD | LTT462 400 mg QD | LTT462 450 mg QD | LTT462 600 mg QD | LTT462 150 mg BID | LTT462 200 mg BID
Number analyzed (Participants) | 2 | 3 | 6 | 4 | 8 | 6 | 11 | 4 | 6 | 12
nanogram per milliliter (ng/mL)
  Day 1: number analyzed (Participants) | 2 | 3 | 6 | 4 | 7 | 6 | 10 | 3 | 5 | 12
  Day 1 | 61.3 (55.9) | 134 (38.8) | 218 (230.9) | 494 (126.8) | 717 (127.4) | 1580 (60.8) | 1420 (83.5) | 1280 (47.7) | 598 (83.0) | 575 (73.8)
  Day 15: number analyzed (Participants) | 2 | 3 | 5 | 3 | 6 | 4 | 8 | 2 | 5 | 6
  Day 15 | 139 (29.9) | 938 (82.5) | 707 (69.0) | 972 (92.4) | 1330 (131.9) | 2370 (83.3) | 3470 (49.7) | 1030 (248.8) | 1390 (58.5) | 1510 (108.0)

12. Secondary Outcome: Area Under the Curve From Time Zero to the Last Measurable Concentration Sampling Time (AUClast) of LTT462
Description: AUClast is the area under the curve from time zero to the last measurable concentration sampling time calculated by mass * time *volume^-1
Time Frame: Cycle 1 Days 1, 2, 3, 8, 15 and 16; Cycle 2 day 1 and 15; Cycle 3 Day 1; Cycle 5 Day 1
Population: PAS included of all participants who have at least 1 PK blood sample providing measurable LTT462 and received at least 1 dose of study drug, didn't vomit within 4 hours postdose, had at least 1 primary PK parameter. Here 'N' number of participants analyzed signifies number of participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | LTT462 45 mg QD | LTT462 100 mg QD | LTT462 150 mg QD | LTT462 200 mg QD | LTT462 300 mg QD | LTT462 400 mg QD | LTT462 450 mg QD | LTT462 600 mg QD | LTT462 150 mg BID | LTT462 200 mg BID
Number analyzed (Participants) | 2 | 3 | 6 | 4 | 7 | 6 | 10 | 3 | 5 | 12
hour*nanogram per milliliter (h*ng/mL) | 851 (106.0) | 2260 (30.0) | 3880 (133.6) | 10400 (95.4) | 12800 (157.4) | 23300 (55.5) | 23800 (115.3) | 11800 (64.2) | 9240 (78.3) | 7630 (98.8)

13. Secondary Outcome: The Time to Reach Maximum (Peak) Plasma, Blood, Serum, or Other Body Fluid Drug Concentration (Tmax) After Single Dose Administration of LTT462
Description: Tmax is the time to reach maximum (peak) plasma, blood, serum, or other body fluid drug concentration after single dose administration.
Time Frame: day 1, day 15
Population: PAS included of all participants who have at least 1 PK blood sample providing measurable LTT462 and received at least 1 dose of study drug, didn't vomit within 4 hours postdose, had at least 1 primary PK parameter. Here 'n' number analyzed signifies number of participants who were evaluable at each time point.
Measure: Median (Full Range); unit: hour
Arm/Group | LTT462 45 mg QD | LTT462 100 mg QD | LTT462 150 mg QD | LTT462 200 mg QD | LTT462 300 mg QD | LTT462 400 mg QD | LTT462 450 mg QD | LTT462 600 mg QD | LTT462 150 mg BID | LTT462 200 mg BID
Number analyzed (Participants) | 2 | 3 | 6 | 4 | 8 | 6 | 11 | 4 | 6 | 12
hour
  Day 1: number analyzed (Participants) | 2 | 3 | 6 | 4 | 7 | 6 | 10 | 3 | 5 | 12
  Day 1 | 2.45 [0.967 to 3.93] | 1.98 [0.867 to 24.0] | 3.49 [2.00 to 24.3] | 5.48 [3.00 to 46.4] | 3.08 [2.08 to 48.8] | 3.04 [1.12 to 4.00] | 3.98 [2.42 to 7.77] | 3.95 [2.00 to 4.20] | 2.25 [2.00 to 49.8] | 3.03 [0.467 to 7.78]
  Day 15: number analyzed (Participants) | 2 | 3 | 5 | 3 | 6 | 4 | 8 | 2 | 5 | 6
  Day 15 | 5.93 [4.00 to 7.85] | 4.02 [1.00 to 4.83] | 4.05 [2.13 to 8.00] | 3.00 [2.17 to 3.02] | 2.59 [1.58 to 4.03] | 2.55 [1.87 to 3.15] | 2.98 [1.00 to 7.62] | 5.25 [3.00 to 7.50] | 2.17 [2.05 to 3.15] | 2.18 [2.00 to 4.15]

14. Secondary Outcome: Elimination Half-life (T1/2) of LTT462
Description: T1/2 is the Elimination half-life.
Time Frame: Cycle 1 Days 1, 2, 3, 8, 15 and 16; Cycle 2 day 1 and 15; Cycle 3 Day 1; Cycle 5 Day 1
Population: as for outcome 12
Measure: Median (Full Range); unit: hour
Arm/Group | LTT462 45 mg QD | LTT462 100 mg QD | LTT462 150 mg QD | LTT462 200 mg QD | LTT462 300 mg QD | LTT462 400 mg QD | LTT462 450 mg QD | LTT462 600 mg QD | LTT462 150 mg BID | LTT462 200 mg BID
Number analyzed (Participants) | 1 | 2 | 4 | 2 | 3 | 6 | 7 | 2 | 2 | 9
hour | 27.9 [27.9 to 27.9] | 39.2 [28.8 to 49.5] | 20.8 [13.4 to 24.5] | 16.8 [16.7 to 16.8] | 15.2 [14.9 to 19.6] | 14.0 [12.0 to 18.7] | 17.6 [16.1 to 18.9] | 13.2 [11.8 to 14.5] | 16.2 [13.3 to 19.1] | 17.1 [11.6 to 41.1]

15. Secondary Outcome: The Area Under the Curve Calculated to the End of a Dosing Interval (Tau) at Steady-state (AUCtau) of LTT462
Description: AUCtau is the area under the curve calculated to the end of a dosing interval (tau) at steady-state calculated by formula amount *time * volume^-1
Time Frame: Cycle 1 Days 1, 2, 3, 8, 15 and 16; Cycle 2 day 1 and 15; Cycle 3 Day 1; Cycle 5 Day 1
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | LTT462 45 mg QD | LTT462 100 mg QD | LTT462 150 mg QD | LTT462 200 mg QD | LTT462 300 mg QD | LTT462 400 mg QD | LTT462 450 mg QD | LTT462 600 mg QD | LTT462 150 mg BID | LTT462 200 mg BID
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 5 | 4 | 4 | 1 | 5 | 4
h*ng/mL | 3010 (NA) — Geometric coefficient of variation was not calculated due to single participant in the arm. | 6370 (NA) — Geometric coefficient of variation was not calculated due to single participant in the arm. | 8660 (50.0) | 14600 (96.5) | 13100 (81.6) | 25400 (74.3) | 35400 (94.8) | 6760 (NA) — Geometric coefficient of variation was not calculated due to single participant in the arm. | 11100 (59.5) | 18600 (85.2)

16. Secondary Outcome: Accumulation Ratio (Racc) of LTT462
Description: Racc is the accumulation ratio calculated by AUCtau ratio Day 15 versus Day 1.
Time Frame: Cycle 1 Days 1, 2, 3, 8, 15 and 16; Cycle 2 day 1 and 15; Cycle 3 Day 1; Cycle 5 Day 1
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | LTT462 45 mg QD | LTT462 100 mg QD | LTT462 150 mg QD | LTT462 200 mg QD | LTT462 300 mg QD | LTT462 400 mg QD | LTT462 450 mg QD | LTT462 600 mg QD | LTT462 150 mg BID | LTT462 200 mg BID
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 4 | 4 | 3 | 0 | 4 | 4
Ratio | 3.01 (NA) — Geometric coefficient of variation was not calculated due to single participant in the arm. | 3.35 (NA) — Geometric coefficient of variation was not calculated due to single participant in the arm. | 5.09 (72.7) | 2.74 (46.9) | 1.49 (25.1) | 1.73 (62.4) | 1.44 (73.4) |  | 3.19 (50.2) | 6.89 (84.3)

17. Secondary Outcome: Changes From Baseline in Relative Quantity (RQ) of Dual Specificity Phosphatase 6 (DUSP6) in Tumor Tissue and in Blood
Description: Assessment of Pharmacodynamic (PD) effects of LTT462 in tumor, pre- and post- treatment tumor biopsies were examined for expression of DUSP6. For assessment of PD effects in blood, levels of DUSP6 were measured in blood samples.
Time Frame: Cycle 1 Days 1, 2, 3, 15 and 16
Population: The full analysis set included all participants who had received at least one dose of LTT462.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | LTT462 45 mg QD | LTT462 100 mg QD | LTT462 150 mg QD | LTT462 200 mg QD | LTT462 300 mg QD | LTT462 400 mg QD | LTT462 450 mg QD | LTT462 600 mg QD | LTT462 150 mg BID | LTT462 200 mg BID
Number analyzed (Participants) | 2 | 3 | 6 | 4 | 8 | 6 | 12 | 6 | 6 | 12
Ratio
  Tumor Sample: number analyzed (Participants) | 1 | 2 | 4 | 1 | 4 | 1 | 4 | 1 | 2 | 3
  Tumor Sample | -0.2 (NA) — Standard deviation was not calculated due to single participant in the arm. | 0.8 (1.11) | -1.1 (29.46) | -28.8 (NA) — Standard deviation was not calculated due to single participant in the arm. | -31.0 (31.06) | -56.5 (NA) — Standard deviation was not calculated due to single participant in the arm. | -22.2 (28.67) | -79.9 (NA) — Standard deviation was not calculated due to single participant in the arm. | -61.8 (4.16) | -14.4 (22.27)
  Blood Sample: number analyzed (Participants) | 2 | 3 | 6 | 3 | 8 | 6 | 12 | 6 | 6 | 11
  Blood Sample | -50.8 (6.14) | -66.1 (40.22) | -35.2 (27.33) | -34.7 (22.02) | -42.5 (16.56) | -43.0 (13.67) | -40.1 (9.92) | -40.4 (21.04) | -39.2 (12.98) | -32.9 (18.71)

ADVERSE EVENTS:
Time Frame: Adverse events were evaluated from screening until at least 30 days after the discontinuation of study treatment (Up to 2.8 years)
Description: The Safety Set included all participants who had received at least one dose of LTT462.
Groups:
- LTT462 600 mg QD: Participants received 450 mg LTT462 QD as oral capsules.
- All QD Participants: Participants received 45 to 600 mg LTT462 QD as oral capsules.
- All BID Participants: Participants received 150 and 200 mg LTT462 BID as oral capsules.
Arm/Group | LTT462 45 mg QD | LTT462 100 mg QD | LTT462 150 mg QD | LTT462 200 mg QD | LTT462 300 mg QD | LTT462 400 mg QD | LTT462 450 mg QD | LTT462 600 mg QD | All QD Participants | LTT462 150 mg BID | LTT462 200 mg BID | All BID Participants
All-Cause Mortality (participants affected / at risk) | 1/2 | 0/3 | 0/6 | 0/4 | 2/8 | 1/6 | 1/12 | 1/6 | 6/47 | 1/6 | 0/12 | 1/18
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/3 | 3/6 | 1/4 | 5/8 | 1/6 | 8/12 | 4/6 | 23/47 | 3/6 | 5/12 | 8/18
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3 | 6/6 | 4/4 | 8/8 | 6/6 | 12/12 | 5/6 | 46/47 | 6/6 | 12/12 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LTT462 45 mg QD (N=2) | LTT462 100 mg QD (N=3) | LTT462 150 mg QD (N=6) | LTT462 200 mg QD (N=4) | LTT462 300 mg QD (N=8) | LTT462 400 mg QD (N=6) | LTT462 450 mg QD (N=12) | LTT462 600 mg QD (N=6) | All QD Participants (N=47) | LTT462 150 mg BID (N=6) | LTT462 200 mg BID (N=12) | All BID Participants (N=18)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 5 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Biliary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Glomerulonephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Renal injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LTT462 45 mg QD (N=2) | LTT462 100 mg QD (N=3) | LTT462 150 mg QD (N=6) | LTT462 200 mg QD (N=4) | LTT462 300 mg QD (N=8) | LTT462 400 mg QD (N=6) | LTT462 450 mg QD (N=12) | LTT462 600 mg QD (N=6) | All QD Participants (N=47) | LTT462 150 mg BID (N=6) | LTT462 200 mg BID (N=12) | All BID Participants (N=18)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 3 | 1 | 2 | 3 | 4 | 3 | 18 | 1 | 3 | 4
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 4 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 4 | 0 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cyanosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Chorioretinopathy (Eye disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 1 | 7 | 0 | 2 | 2
Corneal disorder (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cystoid macular oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Detachment of retinal pigment epithelium (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Macular detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Macular oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 2
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 2 | 1 | 3
Retinal pigment epitheliopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 4 | 0 | 3 | 3
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 4 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 2 | 1 | 0 | 6 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 0 | 1 | 1 | 0 | 6 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 2 | 1 | 4 | 4 | 5 | 3 | 22 | 1 | 5 | 6
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 2 | 1 | 4 | 3 | 3 | 4 | 21 | 3 | 4 | 7
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 4 | 3 | 4 | 4 | 19 | 3 | 4 | 7
Asthenia (General disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 5 | 1 | 1 | 2
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 1 | 2 | 0 | 1 | 2 | 8 | 2 | 4 | 6
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Mucosal dryness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Mucosal haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 6 | 0 | 2 | 2
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 4 | 0 | 1 | 1
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pneumobilia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Urostomy complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 2 | 0 | 2 | 0 | 1 | 2 | 9 | 1 | 0 | 1
Ammonia increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 3 | 3
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 2 | 0 | 1 | 1 | 1 | 2 | 10 | 2 | 3 | 5
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 3 | 0 | 0 | 0 | 2 | 1 | 1 | 7 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 2 | 0 | 4 | 0 | 7 | 0 | 3 | 3
Blood creatinine increased (Investigations) | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 2 | 9 | 0 | 2 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 4 | 0 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 2 | 7 | 0 | 2 | 2
Granulocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipase (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 2 | 2
Liver function test (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 3 | 1 | 2 | 3 | 1 | 3 | 14 | 0 | 3 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0
Hyperalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 1
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1 | 2 | 1 | 1 | 0 | 8 | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 4 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 5 | 3 | 1 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 1
Hypotonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Visual field defect (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prostatic calcification (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 4 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 0 | 6 | 0 | 2 | 2
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 0 | 2 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 2 | 2 | 2 | 0 | 8 | 2 | 2 | 4
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 3 | 2 | 5 | 1 | 14 | 4 | 3 | 7
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 3 | 0 | 2 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 4 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0
Pelvic venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Following careful evaluation of the available study data and considering the limited clinical activity observed with LTT462, the decision was made to not open the dose expansion phase of the study and the study was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/45/NCT02711345/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/45/NCT02711345/SAP_001.pdf